CLINICAL TRIAL: NCT06727344
Title: Comparison of Conservative Treatment With Blood Flow Restriction With Standard Management in Total ACL Rupture. "Randomized Clinical Trial"
Brief Title: Conservative Treatment With Blood Flow Restriction in Patients With Total ACL Rupture. "Randomized Clinical Trial"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Responsible Party: Principal Investigator, Alexios Pitsillides, Alexios Pitsillides BSc, MSc, PhD (cand), European University Cyprus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ΕΕΒΚ/ΕΠ/2024/70
Record Dates: First submitted 2024-11-30; First posted 2024-12-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-11

CONDITIONS: ACL; ACL - Anterior Cruciate Ligament Rupture
Keywords: BFR; Blood Flow Restriction; Brace; ACL rupture; ACL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy; Braces

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brace and BFR exercise (Experimental)
  Interventions: Other: Blood Flow Restriction; Other: Brace
- Brace and BFR sham (Sham Comparator)
  Interventions: Other: Brace

INTERVENTIONS:
Other: Blood Flow Restriction — Exercise with restriction of blood flow supply
  Arms: Brace and BFR exercise
Other: Brace — Knee brace to restrict range of motion

SUMMARY:
The goal of this randomised clinical trial is to evaluate the effects of exercise with blood flow restriction (BFR) in patients with a complete anterior cruciate ligament (ACL) rupture.

The main questions it aims to answer are:

1. Does blood flow restriction adds any additional benefits to conservative treatment of the ACL?
2. Does bracing promotes spontaneous healing to the ACL

Researchers will compare bracing and BFR to bracing and sham BFR to see if the intervention provides any additional benefits to the conservative management of this injury.

Participants will:

1. Use a knee brace for 6 weeks with adjustments according to protocol
2. Follow and identical exercise plan with either BFR (intervention group) or BFR sham (control group)
3. Follow a home based exercise program.

DETAILED DESCRIPTION:
Methodological design:

For the purposes of the present study, a double-blind, two-arm randomised clinical trial will be conducted. Participants in the intervention group will undergo and exercise protocol with the use of blood flow restriction (BFR). Participants in control group will follow the same exercise protocol but with sham BFR instead. Both groups will follow the same brace protocol.

Intervention group:

The intervention group will consist of people with a recent ACL tear who meet the eligibility criteria. Participants in this group will follow a splint use protocol. In particular, during the first 3 weeks (phase 1) a splint will be used with the knee immobilised at 90°, non-weight bearing walking with the use of walking aids according to age and mobility. During the 4th and 5th week (phase 2) the range of motion of the splint will be set to 60° to 90° and from 30° to 90° respectively. Walking will remain non-weight bearing. During the 6th week (phase 3) the degree of freedom of the splint will be placed at 0° allowing full flexion but preventing hyperextension of the joint. During this phase, partial bearing is allowed with the use of a walking aid. From the 7th week (phase 4) onwards the splint is removed and walking is done with no loading restrictions.

Regarding the exercise program, participants in this group, during phase 1, will perform isometric quadriceps and hamstring contractions guided by a visual stimulus from an electronic hand dynamometer. The exercise parameters will be 75 repetitions divided into 4 sets (30,15,15,15) at 30% of the 1st maximum of the opposite leg. During phase 2, the exercise protocol is maintained as phase 1 with the only differences that the exercises will be performed at 60 degrees too. Additionally, the "sliding" exercise will be added where the heel is dragged on the bed causing knee flexion as well as the skateboard sliding exercise from a seated position in the allowed range of motion. Exercise parameters remain the same for all exercises as previous phase. In the 3rd phase, single leg squats up to 45° are added. Exercise parameters remain the same. In the 4th phase, the exercise protocol changes. Subjects start at a stationary bike for 5 minutes (without BFR) and the quadriceps and hamstrings isometrics are replaced with resistance exercises for extension and knee flexion. Sliding and single-leg squats are performed at an increased range of flexion (up to 90°) and climbing a 30cm step is added. All exercise parameters remain the same as in the previous phases. During the last phase (5th) gait retraining on a treadmill for 5 minutes and Y balance exercise is added. Both of these exercises will be performed without BFR. The break between sets will be 30 seconds and between exercises 1 minute.

The exercise program of the intervention group will be performed under lower extremity blood flow restriction. Cuff pressure will be reduced during the breaks. The execution speed of the exercises will be 2 seconds of contraction followed by 2 seconds of return. Hold in all isometric exercises will be 3 seconds.

Initial measurements will be taken upon enrollment of participants and will include MRI, Lachman test, arthrometer, strength, swelling, Lysholm scale, Tegner scale, pain (Vas), exercise pain (Vas). By the end of 2nd and 4th week, strength, swelling and pain (Vas) will be reassessed. The final measurements will be taken at the end of the intervention period and will include all the measurements taken initially.

The participants will be given a home-base exercise program through an electronic platform which will provide the possibility of monitoring their compliance. At the same time, through the platform, the correct execution of the exercises will be ensured as all the exercises will be presented with videos and specific exercise parameters.

Control Group:

The control group will perform an identical program of splinting, exercises, home exercises and measurements as the intervention group. The blood flow restriction protocol will be performed in an identical manner to the intervention group, with only difference being that variables setting will be set at a control program (sham).

ELIGIBILITY:
Inclusion Criteria:

* MRI-confirmed complete rupture of ACL. Ability to communicate and read fluently in Greek and be willing to keep their leg immobilised for the required period based on the study protocol.

Exclusion Criteria:

* Heart disease, overweight, diabetes, pregnancy, thrombophilia, atrial fibrillation, heart failure, cancer, use of drugs that may increase blood clotting, use of hormones or contraceptives, any reason for not using BFR e.g., an open wound or serious skin problems and/or allergies to the cuff material.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Strength | Enrolment, week 2 and 4, end of intervention (12 weeks)
  Quadriceps strength using a hand held dynamometer

SECONDARY OUTCOMES:
MRI | Enrolment and end of intervention at 12 weeks
Knee laxity | enrolment and end of intervention at 12 weeks
  Knee arthrometer
Balance | enrolment and end of intervention at 12 weeks
  Star execution test
Swelling | enrolment and end of intervention at 12 weeks
  Knee circumference
Visual analog scale (VAS) | enrolment, week 2 and 4 and end of intervention at 12 weeks
  Visual analog scale for pain measurement. A higher score indicates greater pain intensity 0 indicates no pain while 100 indicates the worst pain.
Lysholm scale | enrolment and end of intervention at 12 weeks
  Lysholm scale: The Lysholm Knee Score is a questionnaire consisting of 8 items. The scale calculates and grades an overall score from 0 to 100 based on 8 domains: squatting, locking, pain, stair climbing, support, instability, and edema. A high score on the Lysholm score list corresponds to a low degree of knee instability.
Patient reported outcome measures | enrolment and end of intervention at 12 weeks
  Tegner scale:
  The TAS is a one-item questionnaire that is scored on an 11-item scale (0 to 10) based on the patient's reported level of activity/work. A level of 0 represents maximum disability while a level of 10 represents elite sports athletes.

CONTACTS AND LOCATIONS:
Locations (1):
- European University Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No
To keep the study double blinded

REFERENCES:
- [Background] Pitsillides A, Stasinopoulos D, Giannakou K. Healing potential of the anterior cruciate ligament in terms of fiber continuity after a complete rupture: A systematic review. J Bodyw Mov Ther. 2021 Oct;28:246-254. doi: 10.1016/j.jbmt.2021.06.003. Epub 2021 Jun 12. PMID 34776148
- [Background] Filbay SR, Dowsett M, Chaker Jomaa M, Rooney J, Sabharwal R, Lucas P, Van Den Heever A, Kazaglis J, Merlino J, Moran M, Allwright M, Kuah DEK, Durie R, Roger G, Cross M, Cross T. Healing of acute anterior cruciate ligament rupture on MRI and outcomes following non-surgical management with the Cross Bracing Protocol. Br J Sports Med. 2023 Dec;57(23):1490-1497. doi: 10.1136/bjsports-2023-106931. Epub 2023 Jun 14. PMID 37316199
- [Derived] Pitsillides A, Constantinou A, Karagiannis C, Giannakou K. Conservative treatment using blood flow restriction and brace in individuals with complete anterior cruciate ligament rupture: protocol for a randomised clinical trial. J Orthop Surg Res. 2025 Dec 1;21(1):10. doi: 10.1186/s13018-025-06285-y. PMID 41327334